CLINICAL TRIAL: NCT01718496
Title: Physiological Mechanisms of Dyspnea Relief and Improved Exercise Tolerance After Treatment With Oral Morphine in Patients With Advanced Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Morphine, Dyspnea, Exercise and COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jean Bourbeau, respirologist, McGill University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2844
Record Dates: First submitted 2012-10-15; First posted 2012-10-31 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: dyspnea; COPD; exercise tolerance; opioids; morphine; single dose oral Morphine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Morphine; Analgesics, Opioid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Active Comparator): Patient with advance COPD who will randomly receive single dose oral Morphine
  Interventions: Drug: Morphine; Drug: Placebo
- Placebo (Placebo Comparator): patient with advanced COPD who will receive Placebo
  Interventions: Drug: Morphine; Drug: Placebo

INTERVENTIONS:
Drug: Morphine — patient with advanced COPD will randomly receive single dose Morphine to assess its effect on dyspnea and exercise tolerance
  Other Names: Opioids
Drug: Placebo — patients with advanced COPD on the other study arm will randomly receive Placebo
  Other Names: 0.9% Sodium chloride

SUMMARY:
The investigators are studying the effect of a single dose Opioid drug (Morphine) on dyspnea and exercise tolerance in COPD patients.

DETAILED DESCRIPTION:
"Dyspnea" refers to the subjective awareness of breathing discomfort that typically accompanies an increase in physical activity, particularly in patients with Chronic Obstructive Pulmonary Disease (COPD). In these patients, the symptom of dyspnea contributes significantly to exercise intolerance and an impoverished health-related quality of life. Alleviating dyspnea and improving functional capacity are, therefore, among the principal goals of COPD management, i.e., response to therapy. Nevertheless, the effective management of dyspnea and exercise intolerance remains an elusive goal for healthcare providers and current strategies aimed at reversing the patients' underlying chronic disease (e.g., bronchodilators, corticosteroids, supplemental oxygen) are only partially successful in this regard. Evidence-based clinical practice guidelines recommend that, under these circumstances, pain-relieving (opioid) medications may be used for the pharmacologic management of refractory dyspnea and activity-limitation in COPD. Indeed, a handful of published studies provide evidence to suggest that single-dose treatment with morphine or dihydrocodeine improves dyspnea and exercise performance by ~20% in patients with COPD. Nevertheless, little information is available on the physiological mechanisms by which opioid drugs contribute to these improvements in such patients. From a clinical management perspective, this information becomes crucial if we are to optimize the management of exertional symptoms in patients with advanced COPD who remain incapacitated by dyspnea, despite receiving optimal care from their healthcare provider for their underlying disease. Therefore, the purpose of the proposed randomized, double-blind, placebo-controlled, cross-over study is (1) to test the hypothesis that single-dose administration of oral morphine sulphate will improve exertional dyspnea and exercise tolerance in patients with advanced COPD and (2) elucidate the physiological underpinnings of these improvements. To this end, we will compare the effects of single-dose administration of oral morphine sulphate (0.1 mg/kg, equivalent to 7.5 mg for an average 75 kg man) and placebo on dyspnea (sensory intensity and affective responses) and exercise endurance time during symptom-limited constant-work-rate cardiopulmonary cycle exercise testing in symptomatic patients with severe-to-very severe COPD. To explore possible physiological mechanisms of symptom relief, we will measure spirometry parameters, plethysmographic lung volumes and plasma morphine concentrations; perform detailed assessments of central neural respiratory motor drive (i.e., diaphragm electromyography), contractile respiratory muscle function (i.e., esophageal, gastric and transdiaphragmatic pressures), operating lung volumes, ventilation, breathing pattern, pulmonary gas exchange and cardio-metabolic function during exercise; and employ a novel multi-dimensional evaluation technique that permits simultaneous measurement of the sensory intensity and affective dimensions of dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* sever or very sever COPD, i.e. post B2 agonist FEV1<50% predicted
* age >= 40 years
* cigarette smoking history > 2 pack yrs
* ever chronic activity-related dyspnea defined by the combination of A BDI focal score <=6, Modified MRC dyspnea scale >=3 and an OCD rating <=50
* no change in medication dosage & frequency in the preceding 6 weeks
* no hospitalization or exacerbation in the preceding 6 weeks

Exclusion Criteria:

* active cardiopulmonary disease other than COPD
* contraindication to Cardiopulmonary exercise testing
* use of daytime oxygen
* exercise-induced oxyhemoglobin desaturation to <80% on room air
* Body mass index <18.5 or >30 kg/m2
* use of antidepressant drugs in the preceding 2 weeks
* use of opioid drugs in the preceding 4 weeks
* partial pressure of carbon dioxide PCo2 of >50 mmHg on capillary blood gas

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
improvement of dyspnea | one hour
improvement of exercise tolerance | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph. D., Principal Investigator — McGill University
Locations (1):
- Montreal Chest Institute, Montreal, Quebec, Canada